CLINICAL TRIAL: NCT03864952
Title: Dental Plaque and Infectious Agents Story)
Brief Title: Infectious Agents Exposure : Archiving in Dental Plaque
Acronym: DIAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0131 (DIAS study)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Infection; Dental Calculus
Keywords: Infection; genomic; dental calculus
MeSH Terms: conditions — Infections; Dental Calculus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — dental calculus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We are studying the possibility of using dental calculus as a reservoir for the genes of an infectious agent that has infected the patient in previous months; as it is done to highlight climate change in ice samples.

DETAILED DESCRIPTION:
From a sample of people who have had a microbiologically well-documented infection, we will study the possibility after genomic amplification to find, three to 12 months after genetic sequences of the infectious agent in the dental calculus of the person. The people will be recruited according to a large panel of infectious agent (gram + and gram bacterium, mycobacteria, parasite, fungus, DNA, RNA or retrovirus) and, of course, the presence of dental calculus.

ELIGIBILITY:
Inclusion Criteria:

* three months before, having been infected with a documented pathogen
* this infection must have been clinically obvious
* the patient must have dental calculus

Exclusion Criteria:

* to be under 18 years old
* to be incapable to consenting
* a tartar removal since the infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients reffering to the Hospital university of Brest (France) 3 to 12 months before the study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-09-04 (Estimated); Study Completion 2019-09-04 (Estimated)

PRIMARY OUTCOMES:
successful detection of pathogen | 3 to 12 months
  detection of infectious agent

CONTACTS AND LOCATIONS:
Overall Officials: Luc de Saint-Martin, MD, Ph, Study Director — University Hopsital of Brest
Locations (1):
- CHRU de Brest, Brest, France